

## Statistical Analysis Plan

NI-0501-05 Protocol number: Title: A multicentre study for the long-term follow-up of HLH patients who received treatment with NI-0501, an anti-interferon gamma monoclonal antibody SAP Author: SAP Version: Version 1.0, 26 March 2021 DocuSigned by: DocuSigned by: Signer Name: Signer Name: Signing Reason: I approve this document Signing Time: 30-Mar-2021 | 9:06:57 AM CEST Signing Reason: I am the author of this document Signing Time: 30-Mar-2021 | 9:23:18 AM EDT Signature Date Signature Date Approval Author

Veristat

## **Table of contents**

| 1 | | Abbreviations and definition of terms | 4 |
|----|-----|--------------------------------------------------|----|
| 2 | ] | Introduction | 6 |
| 3 | , | Study objectives and endpoints | 7 |
| | 3.1 | Study objectives | 7 |
| | 3.2 | Study endpoints | 8 |
| 4 | , | Study methods | 11 |
| | 4.1 | Overall study design and plan | 11 |
| | 4.2 | Selection of study population | 11 |
| | 4.3 | Method of treatment assignment and randomization | 11 |
| 5 | | Sequence of planned analysis | 12 |
| | 5.1 | Interim analyses | 12 |
| | 5.2 | Analyses and reporting | 12 |
| 6 | | Sample size determination | 12 |
| 7 | | Analysis populations | 12 |
| | 7.1 | Protocol deviations | 13 |
| | 7.2 | COVID-19 | 13 |
| 8 | ( | General issues for statistical analysis | 13 |
| | 8.1 | Handling of missing data and outliers | 14 |
| | 8.2 | Multicenter studies | 14 |
| | 8.3 | Multiple comparisons and multiplicity | 14 |
| | 8.4 | Analysis visit windows | 14 |
| | 8.5 | Derived and computed variables | 15 |
| | | 8.5.1 Efficacy variables: Enrolled-04 cohort | 16 |
| | | 8.5.2 Efficacy variables: Enrolled-06 cohort | 18 |
| 9 | ] | Patient disposition | 19 |
| 10 | ] | Demographics and medical history | 19 |
| | 10. | 1 Demographics | 19 |
| | 10. | 2 Medical history | 20 |
| 11 | | Concomitant medication | 20 |
| 12 | ] | Efficacy analyses | 20 |
| | | 12.1.1 Efficacy analyses: Enrolled-04 cohort | 20 |
| | | 12.1.2 Efficacy analyses: Enrolled-06 Cohort | 21 |
| | | 12.1.3 Efficacy analyses: Enrolled-CU cohort | 21 |
| 13 | | Safety analyses | 21 |

| | 13.1 | Drug exposure | . 22 |
|---|---|---|---|
| | 13 | 3.1.1 Enrolled-04 cohort | .22 |
| | 13 | 3.1.2 Enrolled-06 cohort | .22 |
| | 13 | 3.1.3 Enrolled-CU cohort | .22 |
| | 13.2 | Adverse events | . 22 |
| | 13 | 3.2.1 Serious adverse events | .23 |
| | 13 | 3.2.2 Adverse events leading to study drug withdrawal | .24 |
| | 13 | 3.2.3 Deaths | .24 |
| | 13 | 3.2.4 Infections | .24 |
| | 13.3 | Laboratory data | . 24 |
| | 13.4 | Vital signs | . 25 |
| | 13.5 | Physical examination | . 25 |
| | 13.6 | Pharmacokinetic/pharmacodynamic analysis | . 25 |
| | 13.7 | Immunogenicity – anti-drug antibodies (ADAs) | . 25 |
| | 13.8 | Further safety evaluations | . 26 |
| 14 | Cl | nanges to planned analyses | .26 |
| 15 | Ta | ables, listings, and figures | .26 |
| 16 | Re | eferences | .28 |
| 17 | A | ppendix | .29 |
| | 17.1 | Flow diagram for patients who entered Study NI-0501-05 more than once | . 29 |
| | 17.2 | Adverse events classification by system organ class and preferred term for acute and chronic GvHD and graft failure | |
| | 17.3 | Overall response detailed derivation | .31 |
| | 17.4 | Adverse events indicating organ failure by MedDRA preferred term and code | . 34 |
| | 17.5 | Concomitant medications for HSCT conditioning. | .35 |

## 1 Abbreviations and definition of terms

| ADA | Anti-drug antibodies |
|----------|----------------------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse event |
| AKI | Acute Kidney Injury |
| ALT | Alanine aminotransferase |
| AOSD | Adult-onset Still's Disease |
| ARDS | Acute Renal Failure, Unspecified |
| ASA | American statistical association |
| AST | Aspartate aminotransferase |
| ATC | Anatomical therapeutic chemical |
| CNS | Central Nervous System |
| CI | Confidence intervals |
| COVID-19 | Coronavirus disease 2019 |
| CRF | Case report form |
| CSF | Cerebrospinal fluid |
| CSR | Clinical study report |
| CU | Compassionate use |
| CXCL9 | Chemokine (C-X-C Motif) ligand 9 |
| CXCL10 | Chemokine (C-X-C Motif) ligand 10 |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| FDA | Food and Drug Administration |
| G-CSF | Granulocyte colony stimulating factor |
| gGT | Gamma-glutamyl transferase |
| GvHD | Graft versus host disease |
| HLH | Hemophagocytic lymphohistiocytosis |
| HSCT | Hematopoietic stem cell transplantation |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonisation |
| ΙΕΝγ | Interferon gamma |
| LDH | Lactate dehydrogenase |
| LLN | Lower limit of normal |
| MAS | Macrophage activation syndrome |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic resonance imaging |
| PD | Pharmacodynamic |
| pHLH | Primary hemophagocytic lymphohistiocytosis |


| PK | Pharmacokinetic |
|--------|----------------------------------------------|
| PT | Preferred term |
| RSS | Royal Statistical Society |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SAS® | A software system used for data analysis |
| sCD25 | Soluble CD25 (i.e. soluble IL-2 receptor) |
| SD | Standard deviation |
| SDTM | Study data tabulation model |
| sHLH | Secondary hemophagocytic lymphohistiocytosis |
| sJIA | systemic Juvenile Idiopathic Arthritis |
| Sobi | Swedish Orphan Biovitrum |
| SOC | System organ class |
| TEAE | Treatment-emergent adverse event |
| ULN | Upper limit of normal |
| VAS | Visual Analog Scale |
| WBC | White blood cell |
| WHO-DD | World Health Organization Drug Dictionary |


#### 2 Introduction

This statistical analysis plan (SAP) describes the planned analysis and reporting for Sobi AG protocol number NI-0501-05 ("A multicentre study for the long-term follow-up of HLH patients who received treatment with NI-0501, an anti-interferon gamma monoclonal antibody"). This study has been conducted in North America and Europe according to twin protocols (NI-0501-05-P-IND #111015 and NI-0501-05-EudraCT #2012-005753-23), one for each region, both dated 31-Oct-2019 version 4.0.

This long-term follow-up study is being completed to assess the long-term efficacy and safety of emapalumab for the treatment of hemophagocytic lymphohisticocytosis (HLH) in male and female patients who have received at least one dose of emapalumab in the context of a previous emapalumab clinical study, including patients receiving emapalumab under compassionate use (CU). The research name of emapalumab was NI-0501 and both terms are used interchangeably in this document.

The purpose of this SAP is to outline the planned analyses to be completed to support the Clinical Study Report (CSR) for protocol NI-0501-05. The planned analyses identified in this SAP may be included in regulatory submissions and/or future manuscripts. Exploratory analyses not necessarily identified in this SAP may be performed to support the clinical development program. Any post-hoc, or unplanned, analyses not identified in this SAP will be clearly identified in the CSR.

This SAP includes analysis plans for all patients enrolled in the NI-0501-05 follow-up study. These patients are separated into cohorts based on the parent emapalumab clinical study. These cohorts are described below and outlined in Figure 1:

- Enrolled-04: This cohort includes patients previously enrolled in the NI-0501-04 study, a
  phase 2/3 open-label, single arm, multicenter study to assess safety, tolerability,
  pharmacokinetics, and efficacy of intravenous multiple administrations of emapalumab,
  in the treatment of male and female pediatric patients (≤18 years of age at the time of
  HLH diagnosis) with suspected or confirmed primary HLH (pHLH).
- Enrolled-06: This cohort includes patients previously enrolled in the NI-0501-06 study, a pilot, open-label, single arm, multicenter study to evaluate safety, tolerability, pharmacokinetics, and efficacy of intravenous administrations of emapalumab, an anti-interferon gamma (anti-IFNγ) monoclonal antibody, in patients with systemic Juvenile Idiopathic Arthritis (sJIA) or Adult-onset Still's Disease (AOSD) developing Macrophage Activation Syndrome/secondary HLH (MAS/sHLH).
- Enrolled-CU: This cohort includes patients who were treated under CU and not treated
  under either of the above clinical studies (NI-0501-04 or NI-0501-06). Compassionate
  use treatment was granted to pHLH and sHLH patients having exhausted all possible
  treatment options and who could not be enrolled in a clinical study.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA) and International Council for Harmonisation (ICH): Guidance on Statistical Principles in Clinical Trials<sup>1</sup>. All analyses planned


and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association (ASA)<sup>2</sup> and the Royal Statistical Society (RSS)<sup>3</sup>, for statistical practice.

Figure 1 Overview of the patient cohorts in the NI-0501-05 study



Abbreviations: CU = Compassionate use; MAS = Macrophage Activation Syndrome; pHLH = primary Haemophagocytic lymphohistiocytosis; sHLH = secondary Haemophagocytic lymphohistiocytosis.

Note: There are four patients who entered study NI-0501-05 twice and were assigned separate patient IDs upon re-entry into the study (including 1 patient that received a new ID upon transfer to a different study site). Details are included in Appendix 17.1.

## 3 Study objectives and endpoints

#### 3.1 Study objectives

The study objectives for the NI-0501-05 are as follows:

- · To monitor the long-term safety profile of emapalumab
- To assess HLH patients' survival after emapalumab treatment
- To assess duration of response to emapalumab treatment (ie, maintenance of HLH control)
- To assess post-Hematopoietic Stem Cell Transplantation (HSCT) outcome measures, if applicable


- To assess background disease activity, in patients with secondary forms of HLH
- To study the elimination profile of emapalumab
- To evaluate the pharmacodynamic (PD) effects (levels of circulating total interferon gamma [IFNγ], chemokine (C-X-C Motif) ligand 9 [CXCL9], chemokine (C-X-C Motif) ligand 10 [CXCL10])
- To assess the profile of relevant HLH biomarkers, e.g., sCD25 (soluble CD25)
- · To assess the immunogenicity of emapalumab

#### 3.2 Study endpoints

The study objectives and endpoints are presented in Table 1, including an indicator for which cohort will be assessed for each endpoint.

The safety endpoints of this study are the following:

- Incidence, seriousness, intensity, relationship to emapalumab and outcome of adverse events (AEs)
- Evolution over time of vital signs, physical examination, and laboratory values

The efficacy endpoints are the following:

- Duration of Response after completion of emapalumab treatment (assessed according to the definitions set in the parent study, NI-0501-04 or NI-0501-06).
- Survival time up to one-year post-HSCT (including survival to HSCT and survival post-HSCT) or one year after last emapalumab infusion (if transplant is not performed), calculated from the date of last emapalumab infusion.
- Overall survival calculated as time from the date of last emapalumab infusion to the date of death.
- Post-HSCT outcome indices (applicable only to patients who receive HSCT):
  - Engraftment rate, based on the number of patients experiencing primary or secondary graft failure, as reported as an AE
  - Donor chimerism achieved, based on donor chimerism in peripheral blood completed (i.e., doner cells > 95%)
  - Incidence of acute and chronic graft versus host disease (GvHD), based on occurrence of GvHD, as reported as an AE
- Monitoring of background disease activity (applicable only to patients with sHLH), as assessed by a visual analogue scale (VAS) of MAS activity.

The pharmacokinetics (PK) endpoint is:

• The emapalumab elimination profile, as assessed by levels of circulating emapalumab.

The pharmacodynamics (PD) endpoints include:

- Levels of IFNγ total.
- Exploratory PD parameters/disease markers, including sCD25, CXCL9, CXCL10.


The immunogenicity endpoint is:

• Presence of anti-drug antibodies (ADAs).


Table 1 Study Objectives and Endpoints

| Objective | Endpoints | Population <sup>1</sup> |
|---|---|---|
| To monitor the long-term safety profile of emapalumab | Incidence, seriousness, intensity, relationship to emapalumab and outcome of AEs Evolution over time of vital signs, physical examination, and laboratory values | Enrolled-04<br>Enrolled-06<br>Enrolled-CU |
| To assess pHLH patients' survival after emapalumab treatment | Survival time up to one-year post-HSCT (including survival to HSCT and survival post-HSCT) or one year after last emapalumab infusion (if transplant is not performed or planned) calculated from the date of last emapalumab infusion | Enrolled-04 |
| To assess sHLH patients' survival after emapalumab treatment | Overall survival time up to one year after last emapalumab infusion | Enrolled-06 |
| To assess duration of response<br>to emapalumab treatment (ie.<br>maintenance of HLH control) | Duration of Response after completion of emapalumab treatment (assessed according to the definitions set in the parent study) | Enrolled-04<br>Enrolled-06 |
| To assess post-HSCT outcome measures, if applicable | Post-HSCT outcome indices, e.g., engraftment rate, donor chimerism achieved, incidence of acute and chronic Graft versus Host Disease (GvHD) (it applies to patients who receive HSCT) | Enrolled-04 |
| To assess background disease<br>activity, in patients with<br>secondary forms of HLH | Monitoring of background disease activity (applicable only to patients with sHLH) | Enrolled-06 |
| To study the elimination profile emapalumab | Emapalumab elimination profile | Enrolled-04<br>Enrolled-06<br>Enrolled-CU |
| To evaluate the pharmacodynamic (PD) effects (levels of circulating total IFNγ, CXCL9, CXCL10) | IFNγ total Exploratory PD parameters/disease markers such as sCD25, CXCL9, CXCL10 | Enrolled-04<br>Enrolled-06<br>Enrolled-CU |
| To assess the profile of relevant HLH biomarkers, e.g., sCD25 | Exploratory PD parameters/disease markers such as sCD25, CXCL9, CXCL10 | Enrolled-04<br>Enrolled-06<br>Enrolled-CU |
| To assess the immunogenicity of NI-0501 | Presence of ADAs | Enrolled-04<br>Enrolled-06<br>Enrolled-CU |

<sup>1.</sup> Enrolled-04, Enrolled-06, and Enrolled-CU populations are defined in Section 7.

Abbreviations: AE = adverse event; CXCL9 = chemokine (C-X-C Motif) ligand 9; CXCL1 = chemokine (C-X-C Motif) ligand 10; HSCT = hematopoietic stem cell transplantation; PD = pharmacodynamics; sCD25 = soluble CD25 (ie, soluble IL-2 receptor).


#### 4 Study methods

#### 4.1 Overall study design and plan

This is an international multicentre long-term follow-up study of HLH patients who have received at least one dose of emapalumab in the context of a previous emapalumab clinical study in which no long-term follow-up was already planned. Patients who have received emapalumab under CU treatment protocol may also be considered for enrolment, whenever appropriate.

Patients will enter the NI-0501-05 study either after the last emapalumab infusion or at the end of the short-term follow-up in the parent study, depending on the design of the parent study. Given the fact that patients with different forms of HLH (pHLH or sHLH) can be enrolled in this study, the schedule of assessments differs based on HSCT status: patients who underwent or will undergo HSCT vs. patients for whom HSCT is not planned. Only patients with pHLH are considered for HSCT.

Emapalumab treatment can be continued in the NI-0501-05 study, upon the request of the Investigator in case of the need to delay the schedule for HSCT for reasons unrelated to the administration of emapalumab, provided that a favorable benefit/risk has been established for the patient.

The schedule of assessments for patients enrolled in this study is described in the study protocol, Table 1 for patients who underwent or will undergo HSCT and Table 2 for patients for whom HSCT is not planned. Further assessments for patients continuing emapalumab treatment during the study are described in Appendix A of the study protocol.

#### 4.2 Selection of study population

The study population comprises male and female HLH patients who have received at least one dose of emapalumab in a previous emapalumab clinical study in which no long-term follow-up was planned. An Informed Consent Form (ICF) was signed by the patient or the patient's legal representative(s), as applicable, with the assent of patients who are legally capable of providing it. Patients having received emapalumab under CU were also included where appropriate.

There are no exclusion criteria.

#### 4.3 Method of treatment assignment and randomization

Not applicable.


## 5 Sequence of planned analysis

#### 5.1 Interim analyses

As described in the protocol, data collected in this study may be analyzed on multiple occasions as the study proceeds, in order to facilitate the development programme for emapalumab and to optimize the dissemination of information which may help patient care. These analyses were described in the parent study (NI-0501-04) analysis plan (NI-0501-04 SAP V4 03NOV2017; V5 20SEP2019).

### 5.2 Analyses and reporting

Data for this long-term follow-up study is collected in two separate databases: one for Enrolled-04 and Enrolled-CU, and one for Enrolled-06. Data for each study cohort will be presented separately as described in this SAP.

All final, planned analyses identified in the protocol and in this SAP will be performed only after the last patient has completed the study (last patient last visit) for that cohort, and a data review will be held prior to database lock. The SAP will be finalized and signed prior to the first database lock.

Any post-hoc analyses included which were not identified in this SAP, will be clearly identified as such in the relevant section of the CSR.

#### 6 Sample size determination

A formal sample size calculation was not performed for this long-term, follow-up study. The number of patients enrolled in this study is based on the sample size of the parent studies and under CU.

## 7 Analysis populations

The following analysis populations are planned for this study, separated by cohort as described in Section 2:

- Enrolled-04 includes all consented patients who were previously treated in the NI-0501-04 study.
- <u>Enrolled-06</u> includes all consented patients who were previously treated in the NI-0501-06 study.
- <u>Enrolled-CU</u> includes all consented patients who have been previously treated in CU and were not otherwise treated in a clinical study (NI-0501-04 or NI-0501-06).


#### 7.1 Protocol deviations

Protocol deviations are medically reviewed and categorized as major, minor and exception on an ongoing basis. The final log will be confirmed during a data review meeting, which will be conducted prior to database lock for that cohort. Individual major, minor and exception protocol deviations will be listed by patient.

#### 7.2 COVID-19

A coronavirus disease 2019 (COVID-19) continuity plan has been written to mitigate the negative effects of the COVID-19 pandemic on the conduct of this clinical trial, maintain continuity of study delivery, and, most importantly, ensuring patient safety and wellbeing for patients in the NI-0501-05 study.

The impact of COVID-19 on this clinical trial and trial participants will be included in the listings presenting protocol deviations.

## 8 General issues for statistical analysis

Tabulations will be produced for appropriate demographic, baseline, efficacy, PK, PD, and safety parameters.

Continuous data will be summarized using descriptive statistics: n, mean, standard deviation (SD), median, minimum, and maximum, unless otherwise indicated. Minimum and maximum will be presented to the same number of decimal places as the raw data and mean, standard deviation, standard error of the mean and median will be presented to one more decimal place than the raw data.

Categorical data will be summarized using counts and percentages. Percentages will be suppressed when the count is zero, however the category will still be displayed. The denominator for all percentages will be the number of patients within the group of the population of interest, unless otherwise indicated. Percentages will be presented to one decimal place.

Time-to-event data will be summarized using Kaplan-Meier methodology using 25th, 50th (median), and 75th percentiles with associated 2-sided 95% confidence intervals (CIs), as well as count and percentage of events and censored observations. Endpoints based on binary outcomes, including post-HSCT outcome efficacy measures, will be converted to proportions and associated 95% CIs calculated.

All data will be listed in individual patient data listings. Dates will include a relative study day, presenting the number of days from enrollment (ie, date of consent) in the NI-0501-05 study. Select dates will include a study day, presenting the number of days from date of first dose in the parent study.

Data for each study cohort will be presented separately. For the Enrolled-CU cohort, only listings will be presented, data will not be further summarized in any tables or figures.


Statistical analyses will be performed using SAS software Version 9.4 or later (SAS Institute Inc, Cary, North Carolina, United States).

The immortal time is when subjects cannot experience an event of interest during some period of follow-up time, which can lead to bias if not adequately analyzed. In this study the immortal time is the period between the date of the last visit in the parent study and the date of enrollment in the NI-0501-05 study, thus there is no immortal time for these cohorts by study design.

### 8.1 Handling of missing data and outliers

There will be no imputation for missing or partial dates for AEs or concomitant medications.

For the duration of response efficacy endpoint, imputation methods for missing parameters in assessment of response are described in Section 8.5.1 for the Enrolled-04 cohort and Section 8.5.2 for the Enrolled-06 cohort.

No other imputations of missing data are planned.

#### 8.2 Multicenter studies

As relatively few patients are included in the study, the study sites will not be taken into account in the analyses, and data for each cohort will be pooled across sites.

#### 8.3 Multiple comparisons and multiplicity

No multiplicity adjustment will be considered, since all analyses are descriptive and no formal hypothesis tests are planned for this long-term, follow-up study.

#### 8.4 Analysis visit windows

All statistical analyses will be based on scheduled or unscheduled visits as collected in the Case Report Form (CRF) or as mapped in the source SDTM (study data tabulation model) data. The first visit in NI-0501-05 study will be labeled as "First study-05 visit."

Further details on the mapping of visit labels from the CRF will be documented in the ADaM (analysis data model) define.XML file.

'Baseline' will be used for the baseline visit in the parent study as defined in Section 8.5. These observations will be integrated from the parent study source data in the analysis datasets. For Enrolled-CU not all parameters were collected, therefore baseline from parent study does not apply.


#### 8.5 Derived and computed variables

The following derived variables will be calculated:

- Age (years) at time of consent for the NI-0501-05 study:
   Age (years) = (Date of Informed consent date of birth+1)/365.25
  - Note: The age variable will be calculated to 1 decimal place, to account for patients less than a year old.
- Baseline: the last observation occurring prior to the first treatment administration of emapalumab from the parent study
  - Note: observations occurring on the same day as first treatment administration
    may be the baseline assessment only if the time of assessment occurs prior to the
    time of treatment. If this cannot be determined, the observation will be assumed to
    have occurred after dosing.
- Change from baseline = value at current time point value at baseline
- Relative day (calculated as study day relative to informed consent in study NI-0501-05) =
   Event date date of informed consent +1
- Day (calculated as number of days from the first dose in the parent study) = Event date date of the first dose in the parent study + 1
- Patients who completed the NI-0501-05 study = patients that completed the 1 year visit (i.e., 1 year post HSCT or after last emapalumab infusion)
- Pre-conditioning AEs = any AE with an onset date before the start date of conditioning for HSCT\*
- Post-conditioning AEs = any AE with an onset date on or after the start date of
  conditioning for HSCT\*, applicable only to those patients with an HSCT conditioning
  start date. If the patient received HSCT prior to enrollment (either in NI-0501-04 or CU),
  all AEs in the NI-0501-05 study will be considered as having occurred after HSCT
  conditioning.
- Infection: any AEs from the System Organ Class (SOC) 'Infections and infestations'
- Concomitant medication: any medications that are continuing or start after enrollment (i.e., date of informed consent in NI-0501-05). If an end date is missing or the medication is ongoing at the time of study treatment, the medication will be considered concomitant.

\*Note: The start date of conditioning will be derived based on the start date of the first medication administered for HSCT conditioning, as described in Appendix 17.5.

The following conversion factors will be used to convert days into months or years:

- 1 month = 30.4375 days
- 1 year = 365.25 days

Not all patients will receive treatment under the NI-0501-05 protocol. For those who receive treatment, the definitions of drug administration variables are provided in Table 2, and will be derived using the dosing data from the NI-0501-05 study only.


Table 2: Definition of Drug Administration Variables

| Statistics for Exposure (dosing) | NI-0501-04 and CU |
|---|---|
| Duration of dosing (days and weeks) in NI-0501-05 | Last infusion date - first infusion date+1 (days) (Last infusion date - first infusion date+1)/7 (weeks) |
| Cumulative dose per kg in NI-0501-05 study | Sum of total dose per kg administered from first infusion date until last infusion date in the NI-0501-05 study. |
| Average dose frequency (in days) in NI-0501-05 | Duration of dosing (days) / total number of infusions |
| Average dose (mg/kg) per day in NI-0501-05 | Cumulative dose (mg/kg) / duration of dosing (days) |

## 8.5.1 Efficacy variables: Enrolled-04 cohort

Overall response in the Enrolled-04 cohort is defined as achievement of Complete Response, Partial Response, or HLH Improvement. Criteria for the definition of response are presented in Table 3 and are according to the definitions set in the parent study, Study NI-0501-04. A more detailed specification for implementation of these criteria to derive Overall Response is presented in Appendix 17.3.

**Table 3: Definition of Response** 

| Complete Response | Complete Response is adjudicated if: |
|---|---|
| | • No fever = body temperature < 37.5°C |
| | Normal spleen size confirmed by abdominal ultrasound whenever possible |
| | <ul> <li>No cytopenia = Absolute Neutrophil Counts ≥ 1.0x10<sup>9</sup>/L and platelet count<br/>≥ 100x10<sup>9</sup>/L [absence of G-CSF and transfusion support must be documented for<br/>at least 4 days to report no cytopenia]</li> </ul> |
| | <ul> <li>No hyperferritinemia = serum ferritin level is &lt; 2000 μg/L</li> </ul> |
| | No evidence of coagulopathy, i.e., normal D-Dimer and/or normal (> 150 mg/dL) fibrinogen levels |
| | No neurological and CSF abnormalities attributed to HLH |
| | <ul> <li>No sustained worsening of sCD25 (as indicated by at least two consecutives measurements that are &gt; 2-fold higher than baseline)</li> </ul> |
| Partial Response | Partial Response is adjudicated if: |
| | <ul> <li>At least 3 of the HLH clinical and laboratory abnormalities (including Central Nervous System [CNS] abnormalities) meet the above-mentioned criteria for "Complete Response." In the case of "reactivated patients" who enter the study with 3 abnormal HLH features, at least 2 criteria should meet the definition given</li> <li>There is no progression of other aspects of HLH disease pathology (e.g., jaundice,</li> </ul> |
| | liver size, oedema, CNS clinical alterations) |
| HLH improvement | <ul> <li>Normalization or Improvement (&gt;50% change from baseline) of at least 3 HLH clinical and laboratory abnormalities (including CNS involvement). In the case of "reactivated patients" who enter the study with 2 abnormal HLH features, a change from baseline greater than 50% for both will define HLH as improved.</li> </ul> |


Abbreviations: CSF = cerebrospinal fluid; CNS = central nervous system; HLH = hemophagocytic lymphohistiocytosis; G-CSF = granulocyte colony stimulating factor; sCD25 = soluble CD25 (ie, soluble IL-2 receptor).

For defining Overall Response, values of some parameters may be missing, thus impacting the response assessment. Imputation rules for assessing disease response throughout the study have been pre-defined as follows:

- For calculation of duration of response, both scheduled and unscheduled visits will be used for assessment of response.
- If a parameter needed for the response assessment is missing, the midpoint approach will be used to estimate the missing value i.e., the last observed value before the missing period will be averaged with the first value available after the missing period. Imputed values will be flagged in the listings. This rule will be applied to parameter values missing for a period of up to a maximum of 7 consecutive days. In case that, after imputation, data is still missing in any of the criteria considered for the definition of response, a Complete Response cannot be adjudicated.
- Since data relevant to CNS assessment has been collected at irregular time-points (based on individual patient conditions), the most recent experts' assessment of CNS status will be carried-forward for subsequent time-points.

Cumulative duration of response will be calculated as follows:

- The time in response will be calculated from the first achievement of an Overall Response until start of HSCT conditioning (or end of treatment if the patient did not have HSCT performed). Considering patients may achieve a response, lose that response, and then achieve it subsequently, the total time in response will be calculated by adding together these separate periods in response. Patients who are in response at the time of HSCT conditioning start will be censored at that date. Patients who do not achieve response at least once between the date of first dose and the time of conditioning start are excluded from the analysis.
- Each response duration is defined as the total elapsed time from achievement of response
  to subsequent loss of response, pending the duration of each is at least 4 days. If the
  observed response or loss of response does not last for at least 4 days, then the next
  response period will be considered.
- The start date of conditioning is derived based on the start date of the first medication administered for HSCT conditioning, as described in Appendix 17.5.
- The percentage of days in response will be derived as cumulative response duration divided by number of days from first infusion until HSCT conditioning (or end of treatment if the patient did not have HSCT performed).

#### Survival:

Survival up to HSCT, up to one year post HSCT, and overall survival will be calculated for the Enrolled-04 cohort as follows:


Survival pre HSCT is defined as the time from the date of last dose to the date of death.

Time to death = date of death - date of last emapalumab infusion + 1

Patients who receive an HSCT will be censored at that date. Patients who did not receive HSCT will be censored at last of contact date or 365 days after last dose (whichever comes first).

Survival post HSCT is defined as the time from the date of HSCT (the last HSCT if a
patient has more than one HSCT) to the date of death.

Time to death = date of death - date of HSCT + 1

Patients without an event will be censored at last of contact date or 365 days after last dose (whichever comes first).

Patients who do not proceed to HSCT will be excluded from this analysis.

Overall survival is defined as time from the date of last dose to the date of death. Patients
without an event will be censored the time of last contact or 365 days after last dose
(whichever comes first).

#### 8.5.2 Efficacy variables: Enrolled-06 cohort

Response and duration of response will be derived for the Enrolled-06 cohort as follows:

- Response (MAS remission) after completion of emapalumab treatment (assessed according to the definitions set in the parent study NI-0501-06 (NI-0501-06 SAP V2.0 29OCT20 Section 6.1.7 Derived variables).
  - MAS remission = resolution of clinical signs and symptoms according to the Investigator (defined as a MAS clinical signs and symptoms score  $\leq 1$ ) AND normalization of laboratory parameter relevant to MAS as follows:
    - White blood cell count (WBC) and platelet count above the lower limit of normal (LLN)
    - o Lactate dehydrogenase (LDH) below 1.5 times the upper limit of normal (ULN)
    - Alanine aminotransferase/aspartate aminotransferase (ALT/AST) below 1.5×ULN
    - o Fibrogen higher than 100 mg/dL
    - Ferritin level decreased by at least 80% from values at screening or baseline (whichever is higher) or below 2000 ng/mL, whichever is lower

If one or more laboratory data are unavailable, MAS remission cannot be evaluated.

MAS recurrence is defined as not meeting the above criteria for remission.
 Duration of response will be calculated in the subgroup of patient showing MAS remission during the parent study NI-0501-06, defined as the time from date of first MAS remission during the parent study until the first date of MAS recurrence or death.

date of MAS recurrence/death – date of first MAS remission + 1


Patients who meet the criteria of MAS remission at the end of the study will be censored at the date of last disease assessment (ie, date last known to be in MAS remission).

The MAS remission evaluation is based on a combination of assessments, including Investigator assessment and laboratory findings. The latest date of assessments, within the visit label, will be used for the calculation of the duration of response.

**Survival:** Overall survival time up to one year after last emapalumab infusion will be calculated as follows:

Time to death = date of death - date of last emapalumab infusion + 1

Patients who survive to the end of the study (i.e., beyond 365 days after date of last infusion) will be censored at the date of last contact or 365 days after last dose (whichever comes first). Patients who withdrew consent will be censored at the date of withdrawal of consent.

#### 9 Patient disposition

A tabulation of patient disposition will be provided for the Enrolled-04 and Enrolled-06 cohorts (presented separately). For each cohort, the number of patients for each of the following categories will be presented:

- Number of patients enrolled (i.e., the enrolled population for that cohort)
- Number of patients who received treatment in the NI-0501-05 study
- Number of patients who completed the NI-0501-05 study
- Number of patients who withdrew from the NI-0501-05 study
- Reason for not completing the NI-0501-05 study

Percentages will be calculated using the number of patients in the enrolled population for that cohort.

All disposition data, including the study completion status and the reason for not completing the study will be listed for all cohorts (Enrolled-04, Enrolled-06, and Enrolled-CU). The date of first and last dose received (in either the parent study or NI-0501-05 study) will also be included in the listings.

A by-patient listing of protocol deviations and relationship to COVID-19, as described in Sections 7.1 and 7.2, will be also presented.

#### 10 Demographics and medical history

### 10.1 Demographics

Summary statistics for age at time of consent in the NI-0501-05 study, sex, and race will be tabulated separately for the Enrolled-04 and Enrolled-06 cohorts. A by-patient listing of age, sex,


and race will be presented for all cohorts (Enrolled-04, Enrolled-06, and Enrolled-CU), including height and weight data at first study 05 visit.

#### 10.2 Medical history

All medical history data will be coded using the latest version of Medical Dictionary for Regulatory Activities (MedDRA) version 23.0. Medical history collected in NI-0501-05 study will be presented in listings only for the Enrolled-04 and Enrolled-CU cohorts.

#### 11 Concomitant medication

All concomitant medications will be coded using World Health Organization drug dictionary (WHO-DD) 2019 version or later.

Concomitant medications will be summarized descriptively by Anatomical Therapeutic Chemical (ATC) level 2 and preferred term (PT) using counts and percentages for the Enrolled-04 and Enrolled-06 cohorts.

Any medications that are continuing or start after the enrollment will be considered concomitant. If an end date is missing or the medication is ongoing at the time of study treatment, the medication will be considered concomitant.

Concomitant medications and procedures (including transfusions) will be presented in listings for all cohorts, including a flag for HSCT conditioning medications as applicable. A separate listing for HSCT procedures will be presented for the Enrolled-04 and Enrolled-CU cohorts only.

#### 12 Efficacy analyses

#### 12.1.1 Efficacy analyses: Enrolled-04 cohort

Cumulative duration of response will be presented using descriptive statistics, both overall and as a percentage of days in response.

The survival endpoints (overall survival, survival pre HSCT, and survival post HSCT) will be analyzed descriptively using Kaplan-Meier methodology. The 25th, 50th (median), and 75th percentiles with associated 2-sided 95% CIs, Month 3, 100 days, Month 6, and Month 12 survival probability estimates with associated 95% CIs, as well as count and percentage of events and censored observations will be summarized. A Kaplan-Meier curve will also be presented for each time-to-event endpoint.


#### Binary endpoints:

- Post HSCT engraftment rates: based on the number of patients experiencing primary or secondary graft failure, as reported in the AE module of eCRF (electronic CRF), Appendix 17.1.
- **Post HSCT acute and chronic GvHD incidence:** based on occurrence of GvHD, as reported in the AE module of eCRF, Appendix 17.2.
- **Donor chimerism:** based on donor chimerism in peripheral blood completed (ie, donor cells > 95%) as reported in Chimerism Update module of eCRF.

For these binary secondary endpoints, the number and proportion of patients will be provided with two-sided 95% CIs.

All efficacy data will be provided in data listings.

#### 12.1.2 Efficacy analyses: Enrolled-06 Cohort

The numeric level of background disease activity will be tabulated using descriptive statistics by visit. MAS activity is monitored using a VAS ranging from 0 to 10 by steps of 0.5 (as collected on the CRF).

Duration of response and overall survival will be analyzed descriptively using Kaplan-Meier methodology. The 25th, 50th (median), and 75th percentiles with associated 2-sided 95% CIs, Month 3, 100 days, Month 6, and Month 12 survival probability estimates with associated 95% CIs, as well as count and percentage of events and censored observations will be summarized. A Kaplan–Meier curve will also be presented for each time-to-event endpoint.

All efficacy data, including the parameters used to derive response over time (with baseline values from the parent NI-0501-06 study), will be provided in data listings.

#### 12.1.3 Efficacy analyses: Enrolled-CU cohort

The survival variable (date os death) in the Enrolled-CU cohort will be listed only.

#### 13 Safety analyses

Safety will be evaluated from reported AEs, clinical laboratory findings, changes in vital signs, 12-lead electrocardiograms (ECGs), physical examination results, and emergence of ADAs.

These analyses will be conducted for the Enrolled-04 and Enrolled-06 cohorts separately, with the data from the Enrolled-CU cohort presented in listings only.


#### 13.1 Drug exposure

Not all patients are expected to receive treatment during this long-term, follow-up study. None of the Enrolled-06 patients will receive treatment during the NI-0501-05 study, thus drug exposure will be presented for the Enrolled-04 and Enrolled-CU cohorts only.

#### 13.1.1 Enrolled-04 cohort

The number of patients who received treatment during the NI-0501-05 study will be summarized. Duration of dosing (in days and weeks), cumulative dose per kg, average dose frequency (in days), and average dose (mg/kg) per day will be summarized for those patients who received treatment, using dosing data from the NI-0501-05 study only.

All dosing data will be provided in a data listing.

#### 13.1.2 Enrolled-06 cohort

Study drug exposure is not applicable during the conduct of the NI-0501-05 study.

#### 13.1.3 Enrolled-CU cohort

All dosing data will be provided in data listings, including the derived variables of duration of dosing (in days and weeks), cumulative dose per kg, average dose frequency (in days), and average dose (mg/kg) per day will be listed for those patients who received treatment, using dosing data from the NI-0501-05 study only.

#### 13.2 Adverse events

All AEs and serious AEs (SAEs) will be coded using MedDRA version 23.0. Summaries will be presented separately for the Enrolled-04 and Enrolled-06 cohorts.

For the Enrolled-04 and Enrolled-CU cohorts, AEs will be flagged as occurring pre- or post-HSCT conditioning start, as defined in Section 8.5.

A summary table will present the number and percent of patients reporting as least one of the following:

- AE (overall and by maximum severity)
- Treatment-related AE
- Serious AE
- Treatment-related serious AE
- AE resulting in death


- AE leading to study drug withdrawal (Enrolled-04 and Enrolled-CU cohorts only)
- AE classified as an infection

For the Enrolled-04 cohort, this summary table will be presented for those events occurring pre-HSCT conditioning, post-HSCT conditioning, and overall.

Summaries of the incidence of AEs will be displayed by:

- System Organ Class (SOC) and Preferred Term (PT)
- SOC, PT and maximum severity
- · SOC, PT and maximum relationship to study drug

The AE tables will summarize the incidence of AEs and the number of patients with at least one given AE (sorted in descending order of the total frequency count), including the number of overall events, unless otherwise indicated.

In the case of multiple occurrences of the same AE in the same patient, each patient will only be counted once for each PT. However, all multiple occurrences will be included in the number of events.

In the summary tables by severity and relationship to study drug, the event with the maximum severity or strongest relationship will be reported. If a particular event is missing the severity and/or relationship, then the strongest possible severity or relationship will be assumed for analysis (severity = severe, relationship = related).

By-patient AE data listings with all AEs will be generated.

#### 13.2.1 Serious adverse events

SAEs will be tabulated by:

- SOC and PT
- SOC, PT and maximum severity
- SOC, PT and maximum relationship to study drug

SAEs will be described in a separate data listing.


#### 13.2.2 Adverse events leading to study drug withdrawal

AEs leading to study drug withdrawal will be tabulated by SOC and PT for Enrolled-04 cohort. By-patient data listings of AEs leading to withdrawal will be provided for both Enrolled-04 and Enrolled-CU cohorts.

#### 13.2.3 **Deaths**

By-patient data listings of AEs with a fatal outcome will be displayed.

#### 13.2.4 Infections

AEs classified as an infection will be tabulated by:

PT and maximum severity

All events from the SOC "Infections and infestations" will be presented.

A by-patient listing of all infections reported in the infections log (including search for infections and pathogen details) will be displayed with date of sampling, test, specimen, and result.

#### 13.3 Laboratory data

Shift tables will present changes from baseline (as defined in Section 8.5) to worst on-study and last on-study values relative to normal ranges (ie, below, within, above, or missing) for each parameter, except for ALT, AST, gamma-glutamyl transferase (gGT), LDH, and total bilirubin for which a medically relevant multiple of ULN will be presented. The worst on-study values will be presented by highest and lowest values. For ALT, AST, and gGT medically relevant multiples are 2.5xULN, for LDH and total bilirubin medically relevant multiples are 1.5xULN. Missing categories will be included.

Clinical chemistry, hematology, and coagulation results will be presented in separate tables for the Enrolled-04 and Enrolled-06 cohorts.

Urinalysis results will not be tabulated. Abnormalities in urinalysis results assessed as medically relevant will be recorded as AEs and analyzed as described in Section 13.2.

All laboratory values (including individual change from baseline for Enrolled-04 and Enrolled-06 cohorts) will be displayed in the data listings, including cerebrospinal fluid and pregnancy test results, and those that are outside the normal range will be flagged. A separate listing of all abnormal laboratory results will be presented for all cohorts. Data listings will include both standard and original units.


#### 13.4 Vital signs

Descriptive summaries of actual values by visit will be presented for systolic blood pressure (mmHg), diastolic blood pressure (mmHg), heart rate (bpm), respiratory rate, and highest daily body temperature (Celsius) for Enrolled-04 and Enrolled-06 cohorts.

All vital signs will be provided in data listings for all cohorts.

#### 13.5 Physical examination

By-patient listing of all physical exam data will be displayed by body system: skin, ears/nose/throat, lymphadenopathies, abdominal examination (other than hepato-/spleno-megaly), hepatomegaly, respiratory, cardiovascular, neurological, and other.

Abnormalities related to physical examination and reported as adverse event will be analyzed as described in Section 13.2.

#### 13.6 Pharmacokinetic/pharmacodynamic analysis

PK and PK/PD analyses will be conducted separately and are not included in this SAP.

However, descriptive summaries for the following parameters will be presented by visit (observed results and change from baseline):

- Levels of circulating emapalumab.
- Levels of circulating IFNγ, main IFNγ-induced chemokines (CXCL9, CXCL10), other potential disease markers (sCD25).

Even when no emapalumab was administered within the NI-0501-05 study, PK and PD samples were collected during the study.

These PK/PD will be presented in data listings.

In addition, population PK analysis is planned to be conducted based on the pooled data from Study NI-0501-04, Study NI-0501-05, Study NI-0501-06 and patients treated under CU. Explorative analysis on the relation between emapalumab concentrations and safety parameters may also be conducted. These analyses will be described in a separate data analysis plan.

#### 13.7 Immunogenicity – anti-drug antibodies (ADAs)

A list of patients who developed ADAs will be presented for each cohort.


#### 13.8 Further safety evaluations

Other analyses of safety data, including summaries for different subsets of patients, may be conducted. Any unplanned exploratory analysis performed will be identified as such and described in the final CSR.

The following additional safety data will be included in by-patient listings only:

- 12-lead Electrocardiogram (ECG) results
- Imaging: abdominal ultrasound, chest X-ray, and magnetic resonance imaging (MRI)
  data
- · Hospitalization details

#### 14 Changes to planned analyses

A summary of the changes with respect to analyses described in the study protocol is given below:

- Duration of Response: The protocol (Section 6) states that duration of response after completion of emapalumab treatment will be evaluated. This SAP describes assessment of response throughout the course of participation (either in the parent study or this extension protocol) as follows:
  - Duration of Response for the Enrolled-04 cohort is defined as cumulative response duration, ie, the total number of days in response from the first achievement of response until HSCT conditioning or last treatment date if the patient did not have HSCT performed.
  - Duration of Response for the Enrolled-06 cohort is defined as the number of days between first date of response and first date of loss of response.
- Handling missing data: The protocol (Section 10) stated no imputation of missing data will be applied. In this SAP, for the duration of response efficacy endpoint, imputation methods for missing parameters in assessment of response are described in Section 8.5.1 for the Enrolled-04 cohort and Section 8.5.2 for the Enrolled-06 cohort.

#### 15 Tables, listings, and figures

Table and listing shells are provided as a separate document. No shells are provided for figures.

All tables, listings, and graphs will have a header showing the sponsor company name and protocol and a footer showing the SAS file name and path, and the source of the data (ie, listing number).

The final statistical tables will be produced in the format of the shells and will additionally include "double" page numbering in the format "page xx of yy." The first page numbering ('xx')


will count all pages of the document continuously and the second numbering ('yy') will count the pages for each table separately.

All output will be incorporated into Microsoft Word, or Adobe Acrobat PDF files, sorted and labeled according to the ICH recommendations, and formatted to the appropriate page size(s).


#### 16 References

- US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 2. ASA. (2016) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2016. http://www.amstat.org/about/ethicalguidelines.cfm
- RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf


## 17 Appendix

## 17.1 Flow diagram for patients who entered Study NI-0501-05 more than once

| Patient ID for | Temporal Course of Study Participation | | | |
|---|---|---|---|---|
| Analysis<br>(enrolled cohort) | 1 | 2 | 3 | 4 |
| | NI-0501-04 | NI-0501-05 | CU_NI-0501 | NI-0501-05 |
| (04 cohort) | (pt ID | (pt ID | (pt ID | (pt ID |
| | NI-0501-04 | NI-0501-05 | CU_NI-0501 | NI-0501-05 |
| (04 cohort) | (pt ID | (pt ID | (pt ID | (pt ID |
| | NI-0501-04 | NI-0501-05 | NI-0501-05 | N/A |
| (04 cohort) | (pt ID | (pt ID | (pt ID | |
| | CU_NI-0501 | NI-0501-05 | CU_NI-0501 | N/A |
| (CU cohort) | (pt ID | (pt ID | (pt ID | |


# 17.2 Adverse events classification by system organ class and preferred term for acute and chronic GvHD and graft failure

| System<br>Organ | Contact Contact Class | Preferred<br>Term | Desfermed Towns |
|---|---|---|---|
| Class Code | System Organ Class Chronic GvHD | Code | Preferred Term |
| Acute and C | monic GvIID | | |
| 10021428 | Immune system disorders | 10066264 | Acute graft versus host disease in intestine |
| | | | Acute graft versus host disease in |
| 10021428 | Immune system disorders | 10066262 | skin |
| 10021428 | Immune system disorders | 10018651 | Graft versus host disease |
| | | | Graft versus host disease in |
| 10021428 | Immune system disorders | 10075160 | gastrointestinal tract |
| 10021428 | Immune system disorders | 10064676 | Graft versus host disease in liver |
| 10021428 | Immune system disorders | 10064675 | Graft versus host disease in skin |
| 10021428 | Immune system disorders | 10051396 | Engraftment syndrome |
| Graft Failui | ·e | | |
| | Injury, poisoning and | | |
| 10022117 | procedural complications | 10059032 | Blood stem cell transplant failure |
| | Injury, poisoning and | | |
| 10022117 | procedural complications | 10068081 | Engraft failure |
| | Injury, poisoning and | | |
| 10022117 | procedural complications | 10074860 | Transplant dysfunction |


## 17.3 Overall response detailed derivation

The HLH parameters used to assess disease response for the Enrolled-04 cohort, according to the definition of response reported in Table 3, are described in Table 4. Details for deriving the overall response are described in Table 5.

**Table 4: HLH Parameters for Assessment** 

| HLH Parameter | Variables Used for Assessment | Definition of Normalization |
|---|---|---|
| Parameters that are measured for improvement | | |
| 1. Body temperature | SDTM.VS | Below 37.5°C in all measurements performed on that day |
| 2. Spleen as assessed at physical examination | SDTM.PE | Reported as Normal (= 0 cm from costal margin) |
| 3. Absolute Neutrophil<br>Count and G-CSF<br>administration | SDTM.LB; SDTM.CM where<br>ATC code=L03AA | Absolute Neutrophil Count is equal/greater than 1.0 x 109/L, and no G-CSF has been administered in the previous 4 days |
| 4. Platelet count and platelet transfusion | SDTM.LB; SDTM.PR where<br>PRCAT = Transfusions | Platelet count is equal/greater than 100 x 10 <sup>9</sup> /L, and no platelet transfusion administered in the previous 4 days |
| 5. Ferritin | SDTM.LB | Less than 2000 μg/L |
| 6. Fibrinogen and D-dimers | SDTM.LB | Fibrinogen greater than 1.5 g/L OR D-dimers equal/less than 500 ug/L |
| 7. CNS disease<br>involvement, as assessed by<br>medical team | SDTM.FA | CNS disease ='No' or 'Normalized' means Normal and to be used for CR and PR assessment; CNS= 'Improved' is to be used for HLH improvement assessment |
| Parameters that are measure | ed for worsening of disease | |
| HLH Parameter | Variables Used for Assessment | Definition of Worsening |
| sCD25 levels | SDTM.PD, where PARAMCD = 'sIL2RA' | Percent Change from Baseline (for<br>the last two sCD25 data points<br>before assessment) is not > 200% |
| Ongoing AE which indicates presence of organ failure | SDTM.AE, where organ failure is identified by preferred terms selected by the Sobi medical team, listed in Appendix 17.4 | No ongoing AE at time of response assessment |


**Table 5: Derivation of Overall Response** 

| Response | Application of Criteria | Example |
|---|---|---|
| Complete Response | <ul> <li>All HLH parameters that were abnormal at baseline must be normalized</li> <li>All other parameters that were normal at baseline must still meet the definition of normalized</li> <li>No worsening of disease observed, as assessed by presence of ongoing selected AE or worsening of sCD25 levels</li> </ul> | Subject started with 5 abnormal parameters. All 5 improved, and the remaining parameters continue to meet definition of normalized. There are no ongoing AEs that indicate organ failure. |
| Partial Response | <ul> <li>At least 3 of the HLH parameters that were abnormal at baseline must be normalized. The remaining may be the same or worse as baseline (unless 2 or more parameters no longer meet the definition of normality)</li> <li>Note: If 3 parameters were abnormal at baseline, only 2 need to be normalized. If 2 parameters were abnormal at baseline, only 1 needs to be normalized</li> <li>No worsening of disease observed, as assessed by presence of ongoing selected AE or worsening of sCD25 levels</li> </ul> | Subject started with 4 abnormal parameters. Three (3) of the parameters now meet definition of normalized. The fourth is still abnormal. No more than 1 parameter (normal at baseline) crosses the normality threshold. There are no ongoing AEs that indicate organ failure. |


| Response | Application of Criteria | Example |
|---|---|---|
| HLH Improvement | <ul> <li>At least 3 of the HLH parameters that were abnormal at baseline must be normalized or improved (i.e., &gt;=50% change from baseline). The remaining may be the same or worse as baseline (unless 2 or more parameters no longer meet the definition of normality)</li> <li>Note: If 3 parameters were abnormal at baseline, only 2 need to be at least improved. If 2 parameters were abnormal at baseline, only 1 needs to be improved</li> <li>No worsening of disease observed, as assessed by presence of ongoing selected AE or worsening of sCD25 levels</li> <li>Definition of 50% improvement from baseline:</li> <li>Spleen size decreased by 50%, as recorded in cm from costal margin at physical examination.</li> <li>Absolute Neutrophil Count increased by 50%, if G-CSF has not been administered in the previous 4 days</li> <li>Platelet count increased by 50%, if no platelet transfusion has been administered in the previous 4 days</li> <li>Ferritin decreased by 50%</li> <li>Fibrinogen increased by 50% or D-Dimer decreased by 50%</li> <li>CNS= 'Improved'</li> </ul> | Subject started with 4 abnormal parameters. Two (2) of the parameters now meet definition of normalized. The third improved >50%, but is still abnormal. The fourth is still abnormal and did not improve >50%. No more than 1 parameter (normal at baseline) crosses the normality threshold. There are no ongoing AEs that indicate organ failure. |
| No Response | If a subject does not meet the criteria for at least HLH improvement, response is categorized as "No Response" | Subject meets the definition of partial response, but has worsening disease as identified by an ongoing AE indicating organ failure at time of assessment. |

Abbreviations: AE = adverse event; CNS = central nervous system; HLH = hemophagocytic lymphohistiocytosis; G-CSF = granulocyte colony stimulating factor; sCD25 = soluble CD25 (ie. soluble IL-2 receptor).


## 17.4 Adverse events indicating organ failure by MedDRA preferred term and code

| Preferred Term Code | Preferred Term |
|---------------------|-----------------------------------------|
| 10051093 | Cardiopulmonary failure |
| 10038695 | Respiratory failure |
| 10001053 | Acute respiratory failure |
| 10000804 | Acute hepatic failure |
| 10038435 | Renal failure |
| 10077361 | Multiple organ dysfunction syndrome |
| 10010264 | Condition aggravated |
| 10001051 | ARDS (Acute Renal Failure, Unspecified) |
| 10069339 | AKI (Acute Kidney Injury) |


#### 17.5 Concomitant medications for HSCT conditioning

#### HSCT CONDITIONING

#### **Conditioning Agents to Consider [SDTM.CM]**

| ATC Level 4 | Preferred Code | Preferred Text |
|-------------|----------------|------------------------------|
| L01AA | 00021101001 | CYCLOPHOSPHAMIDE |
| | 00006401001 | MELPHALAN |
| L01AB | 00036801001 | BUSULFAN |
| | 00418901001 | TREOSULFAN |
| L01AC | 00053501001 | ТНІОТЕРА |
| L01BB | 02122001001 | CLOFARABINE |
| | 01004601001 | FLUDARABINE |
| | 01004602001 | FLUDARABINE PHOSPHATE |
| L01BC | 00146201001 | CYTARABINE |
| L01CB | 00511901001 | ETOPOSIDE |
| | 00511902001 | ETOPOSIDE PHOSPHATE |
| L01XC | 01402501001 | RITUXIMAB |
| L04AA | | ALEMTUZUMAB |
| | 0.1.0.00.00.1 | ANTITHYMOCYTE IMMUNOGLOBULIN |
| | 01268601001 | ANTITHYMOCYTE IMMUNOGLOBULIN |
| | 00575401001 | (RABBIT) |
| | 00575402001 | ANTILYMPHOCYTE |
| | 02082701001 | IMMUNOGLOBULIN |

#### Then:

#### For Patients with HSCT date [SDTM.PR]

Med Start Date: >=HSCT date – 16 days (med should start not earlier than 16 days before transplant)

and

- Med End Date: <= HSCT date (med end date should be latest date of transplant)</p>
For Patients without HSCT date [SDTM.PR]

- Med with Indication containing: Conditioning

Start of conditioning is the first start date of any of the selected drugs.




#### **Certificate Of Completion**

Envelope Id:

Subject: Please DocuSign: NI-0501-05 Sobi SAP v1.0\_2021-03-26.pdf

Source Envelope:

Document Pages: 35 Certificate Pages: 5

Signatures: 2 Initials: 0

AutoNav: Enabled

Envelopeld Stamping: Disabled

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

Envelope Originator:



#### **Record Tracking**

Status: Original

3/29/2021 4:56:01 PM

Holder:

Location: DocuSign

Sent: 3/29/2021 4:59:56 PM Viewed: 3/30/2021 3:06:09 AM

Signed: 3/30/2021 3:07:19 AM

Sent: 3/29/2021 4:59:56 PM Viewed: 3/30/2021 9:22:59 AM Signed: 3/30/2021 9:23:26 AM

**Timestamp** 

#### Signer Events

Security Level: Email, Account Authentication

(Required)

Signature



Signature Adoption: Pre-selected Style

Signature ID:



With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

Electronic Record and Signature Disclosure: Accepted: 3/30/2021 3:06:09 AM



Veristat

Security Level: Email, Account Authentication

(Required)



Signature Adoption: Pre-selected Style



With Signing Authentication via DocuSign password

With Signing Reasons (on each tab): I am the author of this document

Electronic Record and Signature Disclosure:

Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |

| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 3/29/2021 4:59:56 PM |
| Certified Delivered | Security Checked | 3/30/2021 9:22:59 AM |
| Signing Complete | Security Checked | 3/30/2021 9:23:26 AM |
| Completed | Security Checked | 3/30/2021 9:23:26 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Veristat (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### How to contact Veristat:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to:

#### To advise Veristat of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from Veristat

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Veristat

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to an email to an email to an email in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send
  this Electronic Record and Disclosure to a location where you can print it, for future
  reference and access; and
- Until or unless you notify Veristat as described above, you consent to receive exclusively
  through electronic means all notices, disclosures, authorizations, acknowledgements, and
  other documents that are required to be provided or made available to you by Veristat
  during the course of your relationship with Veristat.